CLINICAL TRIAL: NCT00828750
Title: Clinical Evaluation of Eltrombopag in Chronic Idiopathic Thrombocytopenic Purpura (ITP)-An Extension Study of Eltrombopag in Subjects, With Idiopathic Thrombocytopenic Purpura (ITP), Previously Enrolled in an Eltrombopag Study TRA108109 (NCT00540423)-<Phase III Study>
Brief Title: Clinical Evaluation of Eltrombopag in Chronic Idiopathic Thrombocytopenic Purpura (ITP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111433
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Results first posted 2011-12-01 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2011-10

CONDITIONS: Idiopathic Thrombocytopenic Purpura; Purpura, Thrombocytopenic, Idiopathic
Keywords: eltrombopag; thrombopoietin receptor agonist; ITP; blood platelet
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag

ARMS (1):
- Treatment (Experimental): Eltrombopag oral tablets once daily
  Interventions: Drug: Eltrombopag oral tablets

INTERVENTIONS:
Drug: Eltrombopag oral tablets — Eltrombopag oral tablets once daily
  Other Names: SB-497115-GR oral tablets

SUMMARY:
An open-label, dose-adjustment extension study to evaluate the safety and efficacy of eltrombopag for treatment of subjects with ITP who have previously been enrolled in the eltrombopag trial TRA108109 (NCT00540423).

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed and dated written informed consent.
* Subject (>=20 years) diagnosed with ITP.
* Subject previously enrolled in TRA108109 (NCT00540423) must have completed the treatment and follow-up periods as defined in that protocol.
* Subject has no intercurrent medical event at risk of thrombosis such as thrombophilia.
* Prolongation of prothrombin time and activated partial thromboplastin time (aPTT) must be within 1.2 times the upper limit of the normal range with no history of hypercoagulable state.
* A complete blood count (CBC), within the reference range, with the following exceptions:
* Hemoglobin: patients with haemoglobin level < the lower limit of normal are eligible for inclusion if hemorrhage is present.
* Neutrophil count >= 1,500/L (1.5x10E9/L) is required for inclusion.
* The following clinical chemistries MUST NOT exceed 1.2 times the upper limit of the normal reference range: creatinine, total bilirubin and alkaline phosphatase.
* The following clinical chemistries MUST NOT exceed 2 times the upper limit of the normal reference range: ALT and AST.
* Albumin must be not less than 80% of the lower limit of normal.
* Female subjects must either be:
* of non-childbearing potential (hysterectomy, bilateral oophorectomy, bilateral tubal ligation or post-menopausal > 1 year), or
* of childbearing potential and have a negative pregnancy test and agree to use contraceptive methods specified in the GSK List of Highly Effective Methods for Avoidance of Pregnancy from two weeks prior to administration of study medication, throughout the study, and 28 days after completion or premature discontinuation from the study:
* Reticulocyte count within the reference range or elevated in case of bleeding.

Exclusion Criteria:

* Any severe medical condition (cardiac, hepatic or renal disorder) other than chronic ITP. (Note: "Severe" is defined as >= Grade 3 as a rule according to the "Classification of the Severity of Adverse Experiences (PAB/SD Notification No.80, dated 29 June 1992)
* History of suspected or confirmed arterial or venous thrombosis (e.g., myocardial infarction, deep vein thrombosis) within the last 1 year.
* History of drug/alcohol abuse or dependence within the last 1 year.
* Suspected blood disorder other than ITP.
* Suspected platelet aggregation abnormality.
* Suspected cyclic thrombocytopenia.
* Suspected Evans Syndrome.
* Subjects who met the GSK Liver Stopping Criteria in the previous eltrombopag study TRA108109 (NCT00540423).
* Current or history of HIV infection or hepatitis B virus or hepatitis C virus infections.
* Current malignancy or history of malignancy that was treated with chemotherapy or radiotherapy.
* Female subjects who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period.
* Subjects who are deemed unsuitable for the study by the investigator (or subinvestigator).
* Treatment with an investigational drug within 30 days preceding the first dose of study medication.
* Pre-existing cardiovascular disease, or arrhythmia known to increase the risk of thromboembolic events (e.g. atrial fibrillation).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Japan (5):
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo

REFERENCES:
- [Derived] Katsutani S, Tomiyama Y, Kimura A, Miyakawa Y, Okamoto S, Okoshi Y, Ninomiya H, Kosugi H, Ishii K, Ikeda Y, Hattori T, Katsura K, Kanakura Y. Oral eltrombopag for up to three years is safe and well-tolerated in Japanese patients with previously treated chronic immune thrombocytopenia: an open-label, extension study. Int J Hematol. 2013 Sep;98(3):323-30. doi: 10.1007/s12185-013-1401-1. Epub 2013 Jul 30. PMID 23896965

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study is an open-label, dose-adjustment extension study to evaluate the safety and efficacy of eltrombopag for the treatment of participants with idiopathic thrombocytopenic purpura (ITP) who had previously been enrolled in eltrombopag trial TRA108109 (NCT00540423).
Groups:
- Eltrombopag: Participants took eltrombopag orally once daily in the fasted state at an individualized dose of 12.5 milligrams (mg), 25 mg, 37.5 mg, or 50 mg; the starting dose was the last dose in the prior eltrombopag study, TRA108109 (NCT00540423). Depending on the participant's platelet count (PC) at each visit, a dose modification guideline allowed participants to increase/reduce the dose or interrupt the eltrombopag treatment.
Period: Overall Study
Arm/Group | Eltrombopag
Started | 19
Completed | 15
Not Completed | 4
Not completed — Lack of Efficacy | 3
Not completed — Normal PC Remained While No Treatment | 1

BASELINE CHARACTERISTICS:
Groups:
- Eltrombopag: Participants took eltrombopag orally once daily in the fasted state at an individualized dose of 12.5 milligrams (mg), 25 mg, 37.5 mg, or 50 mg; the starting dose was the last dose in the prior eltrombopag study, TRA108109 (NCT00540423). Depending on the participant's platelet count at each visit, a dose modification guideline allowed participants to increase/reduce the dose or interrupt the eltrombopag treatment.
Arm/Group | Eltrombopag
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.7 (13.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 7
Race/Ethnicity, Customized [Number; unit: participants]
  Asian - Japanese Heritage | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing an Adverse Event (AE) and/or Serious Adverse Event (SAE) Within the Indicated Category
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of a medical product, whether or not related to the product. An SAE is any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or its prolongation, results in disability/incapacity, is a congenital anomaly/birth defect, or is another event considered serious. A drug-related AE is any AE that was judged to have a relationship with the study medication by the investigator. The severity of an AE is based on the investigator's clinical judgment.
Time Frame: From Baseline (Day 1) to last dose of eltrombopag/early withdrawal visit (up to 981 days)
Population: Safety Population (SP): all participants who received at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 19
participants
  AE | 19
  SAE | 6
  Drug-Related AE | 5
  AE Leading to Withdrawal | 0
  SAE Leading to Withdrawal | 0
  Ongoing AE at the End of Study/Withdrawal | 15
  Mild AE | 6
  Moderate AE | 13
  Severe AE | 0

2. Secondary Outcome: Percentage of Participants Achieving a Platelet Count Greater Than or Equal to 50 Giga Unit (10^9) Per Liter (Gi/L) and Less Than or Equal to 400 Gi/L
Description: Platelet counts were measured by blood draw.
Time Frame: Baseline; Weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, 100, 104, 108, 112, 116, 120, 124, 128, 132, and 136; and last visit/early withdrawal visit (up to Day 982)
Population: Full Analysis Set (FAS): all participants with the exception of those who did not receive any dose of study medication and those with no valid measurements of platelet count on therapy. The number of participants analyzed varies by week because some participants prematurely withdrew and the timing of the measurement differs among participants.
Measure: Number; unit: percentage of participants
Groups:
- Eltrombopag: Participants took eltrombopag orally once daily in the fasted state at an individualized dose of 12.5 mg, 25 mg, 37.5 mg, or 50 mg; the starting dose was the last dose in the prior eltrombopag study, TRA108109 (NCT00540423). Depending on the participant's platelet count at each visit, a dose modification guideline allowed participants to increase/reduce the dose or interrupt the eltrombopag treatment.
Arm/Group | Eltrombopag
Number analyzed (Participants) | 19
percentage of participants
  Baseline, n=19 | 5.3
  Week 1, n=19 | 21.1
  Week 2, n=19 | 63.2
  Week 3, n=19 | 78.9
  Week 4, n=19 | 73.7
  Week 8, n=19 | 73.7
  Week 12, n=16 | 68.8
  Week 16, n=17 | 76.5
  Week 20, n=15 | 73.3
  Week 24, n=17 | 82.4
  Week 28, n=16 | 81.3
  Week 32, n=16 | 68.8
  Week 36, n=18 | 66.7
  Week 40, n=17 | 47.1
  Week 44, n=17 | 58.8
  Week 48, n=18 | 83.3
  Week 52, n=16 | 62.5
  Week 56, n=14 | 57.1
  Week 60, n=16 | 50.0
  Week 64, n=14 | 57.1
  Week 68, n=14 | 57.1
  Week 72, n=12 | 50.0
  Week 76, n=12 | 75.0
  Week 80, n=12 | 66.7
  Week 84, n=13 | 69.2
  Week 88, n=12 | 75.0
  Week 92, n=11 | 72.7
  Week 96, n=11 | 54.5
  Week 100, n=13 | 46.2
  Week 104, n=11 | 45.5
  Week 108, n=11 | 72.7
  Week 112, n=7 | 57.1
  Week 116, n=7 | 85.7
  Week 120, n=5 | 40.0
  Week 124, n=6 | 16.7
  Week 128, n=4 | 25.0
  Week 132, n=2 | 50.0
  Week 136, n=1 | 100
  Last Visit/Early Withdrawal Visit, n=19 | 57.9

3. Secondary Outcome: Median Platelet Counts
Description: Platelet counts were measured by blood draw.
Time Frame: as for outcome 2
Population: FAS. The number of participants analyzed varies by week because some participants prematurely withdrew and the timing of the measurement differs among participants.
Measure: Median (Full Range); unit: Gi/L
Arm/Group | Eltrombopag
Number analyzed (Participants) | 19
Gi/L
  Baseline, n=19 | 20.0 [3 to 117]
  Week 1, n=19 | 36.0 [4 to 308]
  Week 2, n=19 | 84.0 [14 to 463]
  Week 3, n=19 | 85.0 [10 to 194]
  Week 4, n=19 | 97.0 [5 to 259]
  Week 8, n=19 | 102.0 [5 to 224]
  Week 12, n=16 | 85.0 [23 to 238]
  Week 16, n=17 | 76.0 [8 to 217]
  Week 20, n=15 | 61.0 [7 to 252]
  Week 24, n=17 | 70.0 [5 to 255]
  Week 28, n=16 | 97.0 [17 to 202]
  Week 32, n=16 | 75.0 [9 to 184]
  Week 36, n=18 | 73.5 [3 to 233]
  Week 40, n=17 | 45.0 [4 to 222]
  Week 44, n=17 | 59.0 [3 to 226]
  Week 48, n=18 | 71.5 [3 to 224]
  Week 52, n=16 | 81.0 [5 to 303]
  Week 56, n=14 | 58.0 [19 to 223]
  Week 60, n=16 | 48.5 [4 to 252]
  Week 64, n=14 | 57.5 [5 to 201]
  Week 68, n=14 | 53.5 [3 to 200]
  Week 72, n=12 | 51.5 [20 to 188]
  Week 76, n=12 | 90.0 [39 to 241]
  Week 80, n=12 | 67.5 [7 to 277]
  Week 84, n=13 | 86.0 [20 to 280]
  Week 88, n=12 | 65.0 [14 to 205]
  Week 92, n=11 | 78.0 [22 to 194]
  Week 96, n=11 | 57.0 [11 to 236]
  Week 100, n=13 | 45.0 [15 to 282]
  Week 104, n=11 | 44.0 [8 to 241]
  Week 108, n=11 | 69.0 [2 to 318]
  Week 112, n=7 | 56.0 [15 to 146]
  Week 116, n=7 | 84.0 [38 to 148]
  Week 120, n=5 | 21.0 [11 to 294]
  Week 124, n=6 | 32.0 [8 to 156]
  Week 128, n=4 | 37.0 [7 to 178]
  Week 132, n=2 | 34.0 [18 to 50]
  Week 136, n=1 | 51.0 [51 to 51]
  Last Visit/Early Withdrawal Visit, n=19 | 75.0 [7 to 314]

4. Secondary Outcome: Percentage of Participants With a Given Maximum Number of Weeks of Continuous Platelet Count Evaluation Greater Than or Equal to 50 Gi/L and Greater Than or Equal to Twice the Baseline Count Categorized by Weeks on Study Medication (Med.)
Description: Maximum continuous week (MCW) is measured as the longest period (weeks) for which a participant continuously maintained platelet counts greater than or equal to 50 Gi/L and greater than or equal to twice the Baseline count.
Time Frame: From Baseline (Day 1) to last dose of eltrombopag/early withdrawal visit (up to 981 days)
Population: FAS. The number of participants analyzed varies by category of weeks on study medication because the duration of study medication differs among participants.
Measure: Number; unit: percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 19
percentage of participants
  Study Med. =<52 weeks (WKS), MCW=0 week (WK), n=2 | 0
  Study Med. =<52 WKS, MCW >=1 WK, n=2 | 100
  Study Med. =<52 WKS, MCW >=4 WKS, n=2 | 100
  Study Med. =<52 WKS, MCW >=7 WKS, n=2 | 50.0
  Study Med. =<52 WKS, MCW >=10 WKS, n=2 | 50.0
  Study Med. =<52 WKS, MCW >=13 WKS, n=2 | 50.0
  Study Med. =<52 WKS, MCW >=16 WKS, n=2 | 50.0
  Study Med. =<52 WKS, MCW >=19 WKS, n=2 | 50.0
  Study Med. =<52 WKS, MCW >=22 WKS, n=2 | 50.0
  Study Med. =<52 WKS, MCW >=25 WKS, n=2 | 50.0
  Study Med. =<52 WKS, MCW >=28 WKS, n=2 | 50.0
  Study Med. =<52 WKS, MCW >=31 WKS, n=2 | 50.0
  Study Med. =<52 WKS, MCW >=34 WKS, n=2 | 50.0
  Study Med. =<52 WKS, MCW >=37 WKS, n=2 | 0
  Study Med. =<52 WKS, MCW >=40 WKS, n=2 | 0
  Study Med. =<52 WKS, MCW >=43 WKS, n=2 | 0
  Study Med. >52 to =<78 WKS, MCW=0 WK, n=1 | 0
  Study Med. >52 to =<78 WKS, MCW >=1 WK, n=1 | 100
  Study Med. >52 to =<78 WKS, MCW >=4 WKS, n=1 | 100
  Study Med. >52 to =<78 WKS, MCW >=7 WKS, n=1 | 100
  Study Med. >52 to =<78 WKS, MCW >=10 WKS, n=1 | 0
  Study Med. >52 to =<78 WKS, MCW >=13 WKS, n=1 | 0
  Study Med. >52 to =<78 WKS, MCW >=16 WKS, n=1 | 0
  Study Med. >52 to =<78 WKS, MCW >=19 WKS, n=1 | 0
  Study Med. >52 to =<78 WKS, MCW >=22 WKS, n=1 | 0
  Study Med. >52 to =<78 WKS, MCW >=25 WKS, n=1 | 0
  Study Med. >52 to =<78 WKS, MCW >=28 WKS, n=1 | 0
  Study Med. >52 to =<78 WKS, MCW >=31 WKS, n=1 | 0
  Study Med. >52 to =<78 WKS, MCW >=34 WKS, n=1 | 0
  Study Med. >52 to =<78 WKS, MCW >=37 WKS, n=1 | 0
  Study Med. >52 to =<78 WKS, MCW >=40 WKS, n=1 | 0
  Study Med. >52 to =<78 WKS, MCW >=43 WKS, n=1 | 0
  Study Med. >52 to =<78 WKS, MCW >=52 WKS, n=1 | 0
  Study Med. >52 to =<78 WKS, MCW >=65 WKS, n=1 | 0
  Study Med. >78 to =<104 WKS, MCW=0 WK, n=1 | 0
  Study Med. >78 to =<104 WKS, MCW >=1 WK, n=1 | 100
  Study Med. >78 to =<104 WKS, MCW >=4 WKS, n=1 | 100
  Study Med. >78 to =<104 WKS, MCW >=7 WKS, n=1 | 100
  Study Med. >78 to =<104 WKS, MCW >=10 WKS, n=1 | 100
  Study Med. >78 to =<104 WKS, MCW >=13 WKS, n=1 | 100
  Study Med. >78 to =<104 WKS, MCW >=16 WKS, n=1 | 100
  Study Med. >78 to =<104 WKS, MCW >=19 WKS, n=1 | 100
  Study Med. >78 to =<104 WKS, MCW >=22 WKS, n=1 | 100
  Study Med. >78 to =<104 WKS, MCW >=25 WKS, n=1 | 100
  Study Med. >78 to =<104 WKS, MCW >=28 WKS, n=1 | 100
  Study Med. >78 to =<104 WKS, MCW >=31 WKS, n=1 | 100
  Study Med. >78 to =<104 WKS, MCW >=34 WKS, n=1 | 100
  Study Med. >78 to =<104 WKS, MCW >=37 WKS, n=1 | 100
  Study Med. >78 to =<104 WKS, MCW >=40 WKS, n=1 | 100
  Study Med. >78 to =<104 WKS, MCW >=43 WKS, n=1 | 0
  Study Med. >78 to =<104 WKS, MCW >=52 WKS, n=1 | 0
  Study Med. >78 to =<104 WKS, MCW >=65 WKS, n=1 | 0
  Study Med. >78 to =<104 WKS, MCW >=78 WKS, n=1 | 0
  Study Med. >104 to =<130 WKS, MCW=0 WK, n=11 | 0
  Study Med. >104 to =<130 WKS, MCW >=1 WK, n=11 | 100
  Study Med. >104 to =<130 WKS, MCW >=4 WKS, n=11 | 90.9
  Study Med. >104 to =<130 WKS, MCW >=7 WKS, n=11 | 90.9
  Study Med. >104 to =<130 WKS, MCW >=10 WKS, n=11 | 90.9
  Study Med. >104 to =<130 WKS, MCW >=13 WKS, n=11 | 90.9
  Study Med. >104 to =<130 WKS, MCW >=16 WKS, n=11 | 81.8
  Study Med. >104 to =<130 WKS, MCW >=19 WKS, n=11 | 63.6
  Study Med. >104 to =<130 WKS, MCW >=22 WKS, n=11 | 54.5
  Study Med. >104 to =<130 WKS, MCW >=25 WKS, n=11 | 45.5
  Study Med. >104 to =<130 WKS, MCW >=28 WKS, n=11 | 45.5
  Study Med. >104 to =<130 WKS, MCW >=31 WKS, n=11 | 36.4
  Study Med. >104 to =<130 WKS, MCW >=34 WKS, n=11 | 36.4
  Study Med. >104 to =<130 WKS, MCW >=37 WKS, n=11 | 18.2
  Study Med. >104 to =<130 WKS, MCW >=40 WKS, n=11 | 18.2
  Study Med. >104 to =<130 WKS, MCW >=43 WKS, n=11 | 18.2
  Study Med. >104 to =<130 WKS, MCW >=52 WKS, n=11 | 18.2
  Study Med. >104 to =<130 WKS, MCW >=65 WKS, n=11 | 9.1
  Study Med. >104 to =<130 WKS, MCW >=78 WKS, n=11 | 9.1
  Study Med. >104 to =<130 WKS, MCW >=91 WKS, n=11 | 9.1
  Study Med. >104 to =<130 WKS, MCW >=104 WKS, n=11 | 0
  Study Med. >104 to =<130 WKS, MCW >=117 WKS, n=6 | 0
  Study Med. >130 WKS, MCW=0 WK, n=4 | 0
  Study Med. >130 WKS, MCW >=1 WK, n=4 | 100
  Study Med. >130 WKS, MCW >=4 WKS, n=4 | 50.0
  Study Med. >130 WKS, MCW >=7 WKS, n=4 | 50.0
  Study Med. >130 WKS, MCW >=10 WKS, n=4 | 50.0
  Study Med. >130 WKS, MCW >=13 WKS, n=4 | 25.0
  Study Med. >130 WKS, MCW >=16 WKS, n=4 | 25.0
  Study Med. >130 WKS, MCW >=19 WKS, n=4 | 25.0
  Study Med. >130 WKS, MCW >=22 WKS, n=4 | 25.0
  Study Med. >130 WKS, MCW >=25 WKS, n=4 | 25.0
  Study Med. >130 WKS, MCW >=28 WKS, n=4 | 25.0
  Study Med. >130 WKS, MCW >=31 WKS, n=4 | 25.0
  Study Med. >130 WKS, MCW >=34 WKS, n=4 | 25.0
  Study Med. >130 WKS, MCW >=37 WKS, n=4 | 25.0
  Study Med. >130 WKS, MCW >=40 WKS, n=4 | 25.0
  Study Med. >130 WKS, MCW >=43 WKS, n=4 | 0
  Study Med. >130 WKS, MCW >=52 WKS, n=4 | 0
  Study Med. >130 WKS, MCW >=65 WKS, n=4 | 0
  Study Med. >130 WKS, MCW >=78 WKS, n=4 | 0
  Study Med. >130 WKS, MCW >=91 WKS, n=4 | 0
  Study Med. >130 WKS, MCW >=104 WKS, n=4 | 0
  Study Med. >130 WKS, MCW >=117 WKS, n=4 | 0
  Total, MCW=0 WK, n=19 | 0
  Total, MCW >=1 WK, n=19 | 100
  Total, MCW >=4 WKS, n=19 | 84.2
  Total, MCW >=7 WKS, n=19 | 78.9
  Total, MCW >=10 WKS, n=19 | 73.7
  Total, MCW >=13 WKS, n=19 | 68.4
  Total, MCW >=16 WKS, n=19 | 63.2
  Total, MCW >=19 WKS, n=19 | 52.6
  Total, MCW >=22 WKS, n=19 | 47.4
  Total, MCW >=25 WKS, n=19 | 42.1
  Total, MCW >=28 WKS, n=19 | 42.1
  Total, MCW >=31 WKS, n=19 | 36.8
  Total, MCW >=34 WKS, n=19 | 36.8
  Total, MCW >=37 WKS, n=19 | 21.1
  Total, MCW >=40 WKS, n=19 | 21.1
  Total, MCW >=43 WKS, n=19 | 10.5
  Total, MCW >=52 WKS, n=17 | 11.8
  Total, MCW >=65 WKS, n=17 | 5.9
  Total, MCW >=78 WKS, n=16 | 6.3
  Total, MCW >=91 WKS, n=15 | 6.7
  Total, MCW >=104 WKS, n=15 | 0
  Total, MCW >=117 WKS, n=10 | 0

5. Secondary Outcome: Median Number of Maximum Continuous Weeks of Maintaining Platelet Counts Greater Than or Equal to 50 Gi/L and Greater Than or Equal to Twice the Baseline Count at Three-Month Intervals
Description: Maximum continuous week is measured as the longest period (weeks) for which a participant continuously maintained platelet counts greater than or equal to 50 Gi/L and greater than or equal to twice the Baseline count.
Time Frame: 3, 6, 9, 12, 15, 18, 21, 24, 27, and 30 months (13, 26, 39, 52, 65, 78, 91, 104, 117, and 130 weeks)
Population: FAS. The number of participants analyzed varies by category of months (weeks) on study medication because the duration of study medication differs among participants.
Measure: Median (Full Range); unit: weeks
Arm/Group | Eltrombopag
Number analyzed (Participants) | 19
weeks
  Total, n=19 | 19.0 [1 to 91]
  3 Months (13 Weeks), n=18 | 5.0 [0 to 11]
  6 Months (26 Weeks), n=19 | 10.0 [0 to 24]
  9 Months (39 Weeks), n=19 | 12.0 [0 to 36]
  12 Months (52 Weeks), n=17 | 14.0 [0 to 36]
  15 Months (65 Weeks), n=17 | 14.0 [0 to 40]
  18 Months (78 Weeks), n=16 | 15.0 [0 to 53]
  21 Months (91 Weeks), n=15 | 14.0 [0 to 64]
  24 Months (104 Weeks), n=15 | 19.0 [0 to 76]
  27 Months (117 Weeks), n=10 | 17.5 [0 to 91]
  30 Months (130 Weeks), n=4 | 7.5 [3 to 40]

6. Secondary Outcome: Percentage of Participants Experiencing Any Bleeding Episode After Dosing With Study Medication
Description: Any bleeding(s) with an onset on or after the start date of study medication was recorded as a bleeding episode(s).
Time Frame: as for outcome 2
Population: FAS. The number of participants analyzed varies by week because some participants prematurely withdrew and the timing of the evaluation differs among participants.
Measure: Number; unit: percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 19
percentage of participants
  Baseline, n=19 | 63
  Week 1, n=19 | 32
  Week 2, n=19 | 21
  Week 3, n=19 | 16
  Week 4, n=19 | 5
  Week 8, n=19 | 11
  Week 12, n=16 | 13
  Week 16, n=17 | 12
  Week 20, n=15 | 40
  Week 24, n=17 | 6
  Week 28, n=16 | 25
  Week 32, n=16 | 19
  Week 36, n=18 | 39
  Week 40, n=17 | 35
  Week 44, n=17 | 24
  Week 48, n=18 | 22
  Week 52, n=16 | 31
  Week 56, n=14 | 29
  Week 60, n=16 | 13
  Week 64, n=14 | 21
  Week 68, n=14 | 29
  Week 72, n=12 | 8
  Week 76, n=12 | 8
  Week 80, n=12 | 25
  Week 84, n=13 | 0
  Week 88, n=12 | 8
  Week 92, n=11 | 9
  Week 96, n=11 | 9
  Week 100, n=13 | 8
  Week 104, n=11 | 27
  Week 108, n=11 | 27
  Week 112, n=7 | 14
  Week 116, n=7 | 0
  Week 120, n=5 | 0
  Week 124, n=6 | 33
  Week 128, n=4 | 25
  Week 132, n=2 | 50
  Week 136, n=1 | 0
  Last Visit/Early Withdrawal, n=19 | 21

7. Secondary Outcome: Percentage of Participants With a Reduction in Use of Baseline Idiopathic Thrombocytopenic Purpura (ITP) Medication
Description: Concomitant ITP medications included drugs such as steroids and immunosuppressive drugs. Reduction of concomitant ITP medication was defined as a reduction in dose and/or frequency of administration.
Time Frame: From Baseline (Day 1) to last dose of eltrombopag/early withdrawal visit (up to 981 days)
Population: FAS. A total of 15 participants who received at least one concomitant ITP medication at Baseline were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 15
percentage of participants | 87

8. Secondary Outcome: Percentage of Participants Initiating Rescue Medication/Treatment During On-Therapy
Description: Rescue therapy included new ITP medication, an increased dose of a concomitant ITP medication from Baseline (B/L), platelet transfusion, and splenectomy.
Time Frame: From Baseline (Day 1) to last dose of eltrombopag/early withdrawal visit (up to 981 days)
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 19
percentage of participants
  Any Rescue Therapy | 21
  New ITP Medication | 11
  Increase in Concomitant ITP Medication from B/L | 11
  Platelet Transfusion | 0
  Splenectomy | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) with an onset on or after the start date of study medication were collected until the end of the study (up to 981 days).
Arm/Group | Eltrombopag
Serious Adverse Events (participants affected / at risk) | 6/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (N=19)
Cataract (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Cystitis-like symptom (Renal and urinary disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (N=19)
Nasopharyngitis (Infections and infestations) | 12
Bronchitis (Infections and infestations) | 3
Cystitis (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Parotitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tinea infection (Infections and infestations) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Abdominal pain lower (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Food poisoning (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastritis atrophic (Gastrointestinal disorders) | 1
Gastritis erosive (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Reflux oesophagitis (Gastrointestinal disorders) | 1
Tongue discolouration (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Cataract (Eye disorders) | 2
Asthenopia (Eye disorders) | 1
Chalazion (Eye disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Conjunctivitis allergic (Eye disorders) | 1
Eye pruritus (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 2
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1
Heat rash (Skin and subcutaneous tissue disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Chest pain (General disorders) | 2
Fatigue (General disorders) | 2
Pyrexia (General disorders) | 2
Chills (General disorders) | 1
Oedema (General disorders) | 1
Headache (Nervous system disorders) | 4
Hypoaesthesia (Nervous system disorders) | 1
Compression fracture (Injury, poisoning and procedural complications) | 2
Excoriation (Injury, poisoning and procedural complications) | 1
Lip injury (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Aspartate aminotransferase increased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Glucose urine present (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Insomnia (Psychiatric disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 3
Hot flush (Vascular disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Metabolic disorder (Metabolism and nutrition disorders) | 1
Genital haemorrhage (Reproductive system and breast disorders) | 1
Uterine prolapse (Reproductive system and breast disorders) | 1
Presbyacusis (Ear and labyrinth disorders) | 1
Lip neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.